CLINICAL TRIAL: NCT05523323
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Clinical Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) to Evaluate the Safety and Efficacy of Pembrolizumab and Lenvatinib as 1L Intervention in a PD-L1 Selected Population of Participants With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) (LEAP-010).
Brief Title: A Study of Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) as First Line (1L) Intervention in a Programmed Cell Death-ligand 1 (PD-L1) Selected Population With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) (MK-7902-010/LEAP-010)-China Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7902-010 China Extension; MK-7902-010 China Extension (Other: MSD); 205240 (Registry Identifier: JAPIC-CTI); LEAP-10 (Other: MSD)
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; pembrolizumab; lenvatinib; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study was unblinded on August 16, 2023
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Lenvatinib (Experimental): Participants receive lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Lenvatinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- Pembrolizumab + Placebo (Active Comparator): Participants receive lenvatinib-matching placebo orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Lenvatinib-matching placebo will be administered until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib, 20 mg (two 10-mg oral capsules) administered QD
  Other Names: E7080; MK-7902; LENVIMA®
  Arms: Pembrolizumab + Lenvatinib
Biological: Pembrolizumab — Pembrolizumab (MK-3475), 200 mg, every 3 weeks (Q3W) by intravenous (IV) infusion for up to 35 3-week cycles
  Other Names: MK-3475; Keytruda®
Drug: Placebo — Lenvatinib-matching placebo, oral capsules, administered once daily (QD)
  Arms: Pembrolizumab + Placebo

SUMMARY:
This is a study of pembrolizumab (MK-3475) with or without lenvatinib (E7080/MK-7902) as a first line intervention in a PD-L1 selected population with participants with recurrent or metastatic head and neck squamous cell carcinoma.

Hypotheses include:

* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).
* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Progression Free Survival (PFS) per RECIST 1.1 as assessed by BICR.
* Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to overall survival (OS).

DETAILED DESCRIPTION:
The MK-7902-010-China Extension Study will include participants previously enrolled in China in the global study for MK-7902-010 (NCT04199104) plus those enrolled during the China extension enrollment period.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of recurrent/metastatic head and neck squamous cell carcinoma (R/M HNSCC) that is considered incurable by local therapies Note: Participants with newly-diagnosed HNSCC must be M1/Stage IV
* Has a primary tumor location of oropharynx, oral cavity, hypopharynx, or larynx Note: Primary tumor site of nasopharynx (any histology) or unknown primary tumor (including p16+ unknown primary) are not eligible

Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed

* Male participants agree to use approved contraception during the treatment period for at least 7 days after the last dose of lenvatinib/placebo, or refrain from heterosexual intercourse during this period
* Female participants are not pregnant or breastfeeding, and are not a woman of childbearing potential (WOCBP), OR are a WOCBP that agrees to use contraception during the treatment period (or 14 days prior to the initiation of study treatment for oral contraception) and for at least 120 days post pembrolizumab, or 30 days post lenvatinib/placebo, whichever occurs last
* Has measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR) Note: Lesions situated in a previously irradiated area are considered measurable if progression has been showed in such lesions
* Participants with oropharyngeal cancer must have results from testing of human papillomavirus (HPV) status
* Has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function

Exclusion Criteria:

* Has any evidence of symptoms or signs of active tumor bleeding within 6 months before randomization
* Has radiographic evidence of major blood vessel invasion/infiltration or tumor demonstrates >90 degree abutment or encasement of a major blood vessel Note: The degree of proximity to major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis after lenvatinib therapy
* Has a history of re-irradiation to any head and neck sites of disease including the cervical, infraclavicular or supraclavicular lymph nodes for head and neck cancer
* Has ulceration and/or fungation of disease onto the skin surface
* Has a history of any contraindication or has a severe hypersensitivity to any components of pembrolizumab (≥Grade 3) or lenvatinib
* Has pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
* Has a history of a gastrointestinal condition or procedure that, in the opinion of the investigator, may affect oral study drug absorption
* Has clinically significant cardiovascular impairment within 12 months of the first dose of study intervention, such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident/transient ischemic attack (TIA)/stroke, cardiac revascularization, or cardiac arrhythmia associated with hemodynamic instability
* Has disease that is suitable for local therapy administered with curative intent
* Had PD within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC
* Has had major surgery within 3 weeks before to first dose of study interventions
* Has difficulty swallowing capsules or ingesting a suspension orally or by a feeding tube
* Has received prior therapy with lenvatinib or pembrolizumab
* Received last dose of systemic therapy for locoregionally advanced disease less than 6 months before signing consent
* Has received prior therapy with an anti-programmed cell death 1 protein (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-programmed cell death ligand 2 (anti PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention
* Has received a live vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention-administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid) is allowed
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy. (e.g., tuberculosis, known viral or bacterial infections, etc.)
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention
* Has had an allogenic tissue/solid organ transplant
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2025-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (28):
- China (28):
  - Anhui Cancer Hospital-Radiology Department ( Site 3333), Hefei, Anhui
  - Beijing Tongren Hospital affiliated to Capital Medical University ( Site 3343), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 3314), Beining, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 3304), Bejiing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 3327), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 3326), Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 3336), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 3338), Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University ( Site 3344), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 3322), Nanning, Guangxi
  - Guizhou Cancer Hospital ( Site 3330), Guiyang, Guizhou
  - The Third Affiliated Hospital of Harbin Medical University ( Site 3302), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 3309), Zhengzhou, Henan
  - Wuhan Union hospital Cancer Center ( Site 3307), Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 3316), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 3311), Changsha, Hunan
  - Xiangya Hospital of Central South University ( Site 3305), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3334), Changsha, Hunan
  - Changzhou Tumor Hospital - Changzhou Fourth People's Hospital ( Site 3339), Changzhou, Jiangsu
  - Jiangxi Cancer Hospital ( Site 3313), Nanchang, Jiangxi
  - Jilin Cancer Hospital ( Site 3310), Changchun, Jilin
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 3328), Xi'an, Shaanxi
  - Shanghai 9th People hospital ( Site 3332), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 3324), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 3300), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 3308), Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital ( Site 3312), Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital ( Site 3303), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 112 Chinese participants were randomized in the China extension study. Of 112 Chinese participants, 57 participants were randomized in the global portion of the MK-7902-010 (NCT04199104) study and 56 participants were randomized in the China extension portion.
Groups:
- Pembrolizumab + Lenvatinib: Participants received lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Per Amendment (AM) 5, (effective date: 16-Aug-2023), participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
- Pembrolizumab + Placebo: Participants received lenvatinib-matching placebo orally once a day (QD) plus pembrolizumab 200 mg by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (approximately 24 months). Per Amendment (AM) 5, (effective date: 16-Aug-2023), participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Started | 61 | 51
Treated | 61 | 50
Completed | 0 | 0
Not Completed | 61 | 51
Not completed — Death | 26 | 21
Not completed — Ongoing participants | 35 | 30

BASELINE CHARACTERISTICS:
Population: All randomized Chinese participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 61 | 51 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (9.4) | 58.4 (11.0) | 59.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 52 | 48 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 56 | 45 | 101
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 61 | 51 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR based on modified RECIST 1.1 were reported.
Time Frame: Up to approximately 33 months
Population: All randomized Chinese participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 61 | 51
Percentage of participants | 39.3 [27.1 to 52.7] | 9.8 [3.3 to 21.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other; p = 0.0002014, Unstratified Miettinen & Nurminen method; One-sided p-value was calculated using the unstratified Miettinen & Nurminen method; Estimate difference = 29.5, 95% CI 2-sided [14.0 to 43.9] — The exact binomial method by Clopper and Pearson was used to generate the estimate difference and the associated 95% confidence intervals (CIs)

2. Primary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 33 months
Population: All randomized Chinese participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 61 | 51
Months | 7.0 [4.1 to 8.7] | 1.5 [1.4 to 1.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other; p = 0.0000037, unstratified Log-rank test; One-sided p-value was calculated using unstratified Log-rank test; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.21 to 0.55] — The unstratified Cox-Regression model with Efron's method of tie handling with treatment as covariate was used to generate Hazard Ratio (HR) and the associated 95%CI

3. Primary Outcome: Overall Survival (OS)
Description: OS was the time from randomization to death due to any cause.
Time Frame: Up to approximately 33 months
Population: All randomized Chinese participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 61 | 51
Months | 10.9 [8.7 to 17.5] | 11.9 [7.4 to 14.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other; p = 0.30933, Unstratified Log-rank test; One-sided p-value was calculated using unstratified Log-rank test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.49 to 1.54] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death.
Time Frame: Up to approximately 33 months
Population: All randomized Chinese participants with a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 24 | 5
Months | 8.3 [4.6 to NA] — NA = Upper limit of 95%CI for DOR could not be reached due to insufficient number of participants with a response. | NA [5.6 to NA] — NA = Median and upper limit of 95%CI for DOR could not be reached due to insufficient number of participants with a response.

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. Number of participants who experienced an AE will be reported.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 52 months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Up to approximately 33 months
Description: All-cause mortality was analyzed in all randomized Chinese participants. Serious and non-serious adverse events (AEs) were reported in all randomized Chinese participants who received at least 1 dose of study treatment. MedDRA 26.0 preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug were excluded. Second course AEs were not reported since no Chinese participants were eligible for second course treatment.
  .
Groups:
- Pembrolizumab + Lenvatinib - First Course: Participants received lenvatinib 20 mg orally once a day (QD) plus pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W). Pembrolizumab will be administered for up to 35 cycles (approximately 24 months). Per Amendment (AM) 5, (effective date: 16-Aug-2023), participants discontinued lenvatinib and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
- Pembrolizumab + Placebo - First Course: Participants received lenvatinib-matching placebo orally once a day (QD) plus pembrolizumab 200 mg by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (approximately 24 months). Per Amendment (AM) 5, (effective date: 16-Aug-2023), participants discontinued placebo and participants who remained on treatment received open-label pembrolizumab only. Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) or who attained complete response (CR) but experienced progression of disease (PD), initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 each 3-week cycle (Q3W), for up to 17 cycles (up to ~1 year).
Arm/Group | Pembrolizumab + Lenvatinib - First Course | Pembrolizumab + Placebo - First Course
All-Cause Mortality (participants affected / at risk) | 26/61 | 21/51
Serious Adverse Events (participants affected / at risk) | 31/61 | 17/50
Other Adverse Events (participants affected / at risk) | 56/61 | 40/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib - First Course (N=61) | Pembrolizumab + Placebo - First Course (N=50)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (5)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Infected metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib - First Course (N=61) | Pembrolizumab + Placebo - First Course (N=50)
Anaemia (Blood and lymphatic system disorders) | 20 (32) | 18 (24)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 5 (6)
Hyperthyroidism (Endocrine disorders) | 4 (7) | 2 (2)
Hypothyroidism (Endocrine disorders) | 34 (41) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (5)
Fatigue (General disorders) | 4 (4) | 3 (3)
Malaise (General disorders) | 7 (7) | 5 (5)
Pyrexia (General disorders) | 7 (7) | 3 (4)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia (Infections and infestations) | 8 (8) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (7) | 8 (10)
Amylase increased (Investigations) | 2 (2) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 9 (13) | 6 (10)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 4 (5)
Blood bilirubin increased (Investigations) | 8 (8) | 1 (1)
Blood creatinine increased (Investigations) | 4 (5) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 7 (7) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (4)
Lipase increased (Investigations) | 4 (4) | 3 (3)
Lymphocyte count decreased (Investigations) | 4 (9) | 2 (3)
Neutrophil count decreased (Investigations) | 5 (11) | 2 (3)
Platelet count decreased (Investigations) | 15 (21) | 4 (4)
Urinary occult blood positive (Investigations) | 5 (11) | 2 (2)
Weight decreased (Investigations) | 21 (23) | 11 (12)
White blood cell count decreased (Investigations) | 8 (15) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (8) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (13) | 9 (9)
Hypochloraemia (Metabolism and nutrition disorders) | 6 (12) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (14) | 8 (10)
Hypoproteinaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 2 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 6 (7)
Haematuria (Renal and urinary disorders) | 6 (10) | 1 (1)
Proteinuria (Renal and urinary disorders) | 24 (43) | 6 (9)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (16) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Hypertension (Vascular disorders) | 32 (59) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT05523323/Prot_SAP_000.pdf